CLINICAL TRIAL: NCT04191915
Title: Assessment of Frailty in Elderly Patients Undergoing Elective Cardiac Surgery
Brief Title: Frailty Assessment in Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital (Other)
Collaborators: Turkish Society of Cardiovascular Surgery (Unknown)
Responsible Party: Principal Investigator, Kamile Ozeren Topcu, Principal Investigator, Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital
Other Study IDs: HNEAH-KAEK 2019/76
Record Dates: First submitted 2019-12-05; First posted 2019-12-10 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Frailty
Keywords: Aged; Cardiac Surgical Procedures; Coronary Artery Disease; Frail Elderly; Frailty; Heart Valve Diseases
MeSH Terms: conditions — Frailty; Coronary Artery Disease; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Frail: Participants with 3 or more components of Fried frailty scale
- Moderately Frail: Participants with 1-2 components of Fried frailty scale
- Not Frail: Participants without any components of Fried frailty scale

SUMMARY:
With increasing life expectancy, cardiac surgical procedures are increasingly being performed in older adults. The biological syndrome of frailty is an aging-associated state with diminished physiological reserve and resistance to stressors, such as major surgery. In the European System for Cardiac Operative risk Evaluation (EuroSCORE II) and the Society of Thoracic Surgeons (STS) risk scoring systems, patient comorbidities including advanced age and poor mobility are considered as risk factors for operative mortality. However, an objective assessment of frailty is not included. Traditionally, frailty assessment before cardiac surgery is primarily performed based on surgeon's subjective perception of patient's general appearance. Objective measurement of frailty is increasingly being applied as a routine part of preoperative evaluation of elderly patients undergoing cardiac surgery. The most widely used frailty assessment tool is the Fried scale. The investigators aim to investigate whether Fried scale would predict operative mortality and morbidity in elderly patients undergoing elective cardiac surgery.

DETAILED DESCRIPTION:
Consecutive patients who are scheduled to undergo elective cardiac surgery in Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital will be evaluated for enrollment. Those who meet inclusion and exclusion criteria will be invited to be study participants. Volunteers will constitute the study population. All participants will undergo routine preoperative risk assessment procedures of our institution, which include history, physical examination, blood chemistry, chest X-ray, echocardiogram, and spirometry. As part of this routine assessment, Fried scale (5-meter walk test, hand-grip strength, questioning of weight loss, short version of the Center for Epidemiological Studies-Depression scale, and short version of the Minnesota Leisure Time Physical Activity questionnaire) will be applied to all participants. Demographics characteristics and clinical data will be observed and recorded. Participants will be divided into 3 groups according to Fried scale; frail, moderately frail, and not frail.

In order to investigate the ability of Fried scale to predict cardiac operative mortality and morbidity, groups will be compared in terms of surgical mortality, renal failure, stroke, prolonged mechanical ventilation, deep sternal wound infections, re-operation, prolonged length of stay, and readmission rates.

Power analysis was performed to estimate sample size using G*Power (v3.1.7) software. A total 150 participants are needed in order to achieve an 80% (Beta=0.2) power at the 5% (Alpha=0.05) level of significance.

Categorical data will be presented as frequency and percentage. Continuous variables will be presented as mean [±standard deviation] and median [interquartile range]. Categorical variables will be compared using chi-square and Fisher's exact tests. Kolmogorov-Smirnov test will be used to assess distribution of continuous variables. Continuous variables with a normal distribution will be compared using Student's t-test, and those with a non-normal distribution will be compared using Mann-Whitney U test.

SPSS for Windows v.17.0 (SPSS Statistics Inc., Chicago, Ill., USA) will be used for all statistical analyses. A two-sided p value of <0.05 will be considered to be statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Age≥65 years
* Planned elective cardiac surgery

Exclusion Criteria:

* Age<65 years
* Emergent procedure
* Refusal to participate
* Clinical instability (recent myocardial infarction, decompensated cardiac failure, acutely symptomatic participants, abnormal vital signs)
* Canadian Cardiovascular Society grade IV angina pectoris
* New York Heart Association class IV heart failure
* Failure to cooperate due to neuropsychiatric disorders

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients scheduled to undergo elective cardiac surgery in Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital
Sampling Method: Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Operative Mortality or Major Morbidity | 30 days
  Composite endpoint defined by The Society of Thoracic Surgeons. Operative mortality is defined as death occurring within 30 days after surgery, or during the same hospitalization following surgery.
  Major morbidity includes permanent stroke, renal failure, prolonged ventilation, deep sternal wound infection, re-operation for any reason.

SECONDARY OUTCOMES:
Number of Participants with Prolonged Length of Stay | 14 days
  Failure to be discharged within 14 days of surgery
Number of Participants with Prolonged Length of Intensive Care Unit Stay | 48 hours
  Length of intensive care unit stay ≥ 48 hours
Number of Participants with Readmission to Intensive Care Unit | 30 days
  Unplanned readmission to intensive care unit during index hospitalization
Number of Participants with Readmission to hospital | 30 days
  Rehospitalization for any reason within 30 days of discharge

CONTACTS AND LOCATIONS:
Overall Officials: Ilyas Kayacioglu, M.D., Study Director — Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital
Locations (1):
- Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Henry L, Halpin L, Barnett SD, Pritchard G, Sarin E, Speir AM. Frailty in the Cardiac Surgical Patient: Comparison of Frailty Tools and Associated Outcomes. Ann Thorac Surg. 2019 Jul;108(1):16-22. doi: 10.1016/j.athoracsur.2019.03.009. Epub 2019 Apr 3. PMID 30953654
- [Background] Rowe R, Iqbal J, Murali-Krishnan R, Sultan A, Orme R, Briffa N, Denvir M, Gunn J. Role of frailty assessment in patients undergoing cardiac interventions. Open Heart. 2014 Feb 1;1(1):e000033. doi: 10.1136/openhrt-2013-000033. eCollection 2014. PMID 25332792
- [Background] Bagnall NM, Faiz O, Darzi A, Athanasiou T. What is the utility of preoperative frailty assessment for risk stratification in cardiac surgery? Interact Cardiovasc Thorac Surg. 2013 Aug;17(2):398-402. doi: 10.1093/icvts/ivt197. Epub 2013 May 10. PMID 23667068
- [Background] Sundermann SH, Dademasch A, Seifert B, Rodriguez Cetina Biefer H, Emmert MY, Walther T, Jacobs S, Mohr FW, Falk V, Starck CT. Frailty is a predictor of short- and mid-term mortality after elective cardiac surgery independently of age. Interact Cardiovasc Thorac Surg. 2014 May;18(5):580-5. doi: 10.1093/icvts/ivu006. Epub 2014 Feb 3. PMID 24497604
- [Background] Sundermann S, Dademasch A, Rastan A, Praetorius J, Rodriguez H, Walther T, Mohr FW, Falk V. One-year follow-up of patients undergoing elective cardiac surgery assessed with the Comprehensive Assessment of Frailty test and its simplified form. Interact Cardiovasc Thorac Surg. 2011 Aug;13(2):119-23; discussion 123. doi: 10.1510/icvts.2010.251884. Epub 2011 Mar 4. PMID 21378017
- [Background] Sundermann S, Dademasch A, Praetorius J, Kempfert J, Dewey T, Falk V, Mohr FW, Walther T. Comprehensive assessment of frailty for elderly high-risk patients undergoing cardiac surgery. Eur J Cardiothorac Surg. 2011 Jan;39(1):33-7. doi: 10.1016/j.ejcts.2010.04.013. PMID 20627611
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Afilalo J, Alexander KP, Mack MJ, Maurer MS, Green P, Allen LA, Popma JJ, Ferrucci L, Forman DE. Frailty assessment in the cardiovascular care of older adults. J Am Coll Cardiol. 2014 Mar 4;63(8):747-62. doi: 10.1016/j.jacc.2013.09.070. Epub 2013 Nov 27. PMID 24291279
- [Background] Singh M, Stewart R, White H. Importance of frailty in patients with cardiovascular disease. Eur Heart J. 2014 Jul;35(26):1726-31. doi: 10.1093/eurheartj/ehu197. Epub 2014 May 26. PMID 24864078
- [Background] Afilalo J, Karunananthan S, Eisenberg MJ, Alexander KP, Bergman H. Role of frailty in patients with cardiovascular disease. Am J Cardiol. 2009 Jun 1;103(11):1616-21. doi: 10.1016/j.amjcard.2009.01.375. Epub 2009 Apr 8. PMID 19463525